CLINICAL TRIAL: NCT05301738
Title: Plyometric Exercise-induced Mechanical and Morphological Changes in Plantar Flexors' Muscle-tendon Unit in Children With Unilateral Cerebral Palsy: A Randomized Controlled Trial
Brief Title: Plyometric Exercise-induced Mechano-morphological Changes of Plantar Flexor Muscle-tendon Unit in Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ragab Kamal Elnaggar, Associate Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RHPT/0020/0059
Record Dates: First submitted 2022-03-20; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Plyometric Exercise

STUDY DESIGN:
Intervention Model Description: A prospective pre-test post-test randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: This was a single-blind protocol. The researcher who collected the data was blind to the allocation of treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plyometric exercise group (Experimental): Participants in this group received the plyometric training program
  Interventions: Other: Plyometric Exercises
- Control group (Active Comparator): Participants in this group received the standard physical rehabilitation program
  Interventions: Other: Standard Physical Therapy

INTERVENTIONS:
Other: Plyometric Exercises — The plyometric exercise group received a 12-week plyometric training program. Each session lasted 45 minutes and was repeated two times a week. The training was conducted in conformity with the National Strength and Conditioning Association guidelines and American Academy of Pediatrics safety standards. The plyometric exercise program consisted of ten unilateral and bilateral lower limb plyometrics in the form of hopping/bounding/jumping activities. The Iplyometric workout was proceeded by a 5-minute warm-up and ended up with a 5-minute cool-down
  Arms: Plyometric exercise group
Other: Standard Physical Therapy — The control group received their usual physical rehabilitation program for 45 minutes, twice/week for 12 consecutive weeks. The program comprised advanced balance training, and gait training exercises, postural and flexibility exercises, strength training exercises.
  Arms: Control group

SUMMARY:
This study was designed to investigate the effect of three months of plyometric exercise training on the mechanical and morphological properties of the plantar flexor muscle-tendon unit in children with unilateral cerebral palsy (UCP). Thirty-eight children with UCP were randomly allocated to the plyometric exercise group (n = 19, underwent a plyometric training program) or the Control group (n =19, received usual physical rehabilitation alone). Both groups were assessed for the plantar flexors' morphological and mechanical properties before and after treatment.

DETAILED DESCRIPTION:
Thirty-eight children with CP participated in the study. They were recruited from King Khalid Hospital and Physical Therapy Center of College of Applied Medical Sciences at Prince Sattam bin Abdulaziz University, Al-Kharj, Saudi Arabia. Their age ranged between 10 and 16 years, were functioning at levels I or II according to the Gross Motor Function Classification System, and had spasticity level 1 or 1+ per the Modified Ashworth Scale. Children were excluded if they had nonreducible structural deformities, received neurolytic agents such as BOTOX or Phenol injections in the past six months, underwent neuromuscular or orthopedic surgery in the last 12 months, or if they had cardiopulmonary problems preventing them from performing high-intense exercise training.

Outcome measures

1. Plantar Flexors' Morphological Properties: length of gastrocnemius muscle-tendon unit, gastrocnemius muscle belly, and achilles, in addition to fascicle length, pennation angle, and gastrocnemius muscle thickness were assessed using a standard high-resolution ultrasound imaging system.
2. Plantar Flexors' Mechanical Properties: Passive range of motion of the ankle joint and maximum isometric voluntary contraction were assessed using an isokinetic dynamometer.

The plyometric exercise group received a 12-week plyometric training program. Each session lasted 45 minutes and was repeated two times a week. The training was conducted in conformity with the National Strength and Conditioning Association guidelines and American Academy of Pediatrics safety standards. The plyometric exercise program consisted of ten unilateral and bilateral lower limb plyometrics in the form of hopping/bounding/jumping activities. The Iplyometric workout was proceeded by a 5-minute warm-up and ended up with a 5-minute cool-down. The control group received their usual physical rehabilitation program for 45 minutes, twice/week for 12 consecutive weeks. The program comprised advanced balance training, and gait training exercises, postural and flexibility exercises, strength training exercises.

ELIGIBILITY:
Inclusion Criteria:

* Hemiparetic cerebral palsy
* Age between 10 to 16 years
* Spasticity level 1 or 1+ according to the Modified Ashworth Scale
* Gross motor function level I or II according to the Gross Motor Function Classification System

Exclusion Criteria:

* Structural deformities
* Musculoskeletal or neural surgery in the last year
* BOTOX injection in the last 6 months.
* Cardiopulmonary disorders limit the ability to engage in explosive exercise training
* Perceptual and behavioral disorders.

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-12-02 (Actual); Study Completion 2021-12-02 (Actual)

PRIMARY OUTCOMES:
Gastrocnemius muscle-tendon length | 2 months
  The distance from the medial femoral epicondyle to the insertion of the Achilles tendon on the calcaneus. The gastrocnemius muscle-tendon length normalized to the lower limb length (%) was recorded.
Achilles tendon length | 2 months
  The distance from the gastrocnemius muscle-tendon junction to its insertion. The achilles tendon length normalized to the lower limb length (%) was recorded.
Gastrocnemius muscle belly length | 2 months
  Distance between the medial femoral epicondyle and its muscle-tendon junction. The gastrocnemius muscle belly length normalized to the lower limb length (%) was recorded.
Fascicle length | 2 months
  The linear distance (mm) between the insertion into the deep and superficial aponeurosis.
Pennation angle | 2 months
  The angle (in degrees) between the fascicle and the deep aponeurosis.
Gastrocnemius muscle thickness | 2 months
  The perpendicular distance (mm) between the deep and superficial aponeurosis.
Passive range of motion of the ankle | 2 months
  The passive ankle dorsi and plantar flexion angle (degrees) were measured by moving the ankle into maximum dorsiflexion and plantarflexion through the isokinetic dynamometry.
Isometric maximum voluntary contractions of the plantar flexors. | 2 months
  The isometric maximum voluntary contraction was determined as the maximum rate of force (Nm) that participants were able to develop during an isometric contraction of the plantar flexors with the ankle in a neutral position (90 degrees) and the knee in a full extension.
Achilles tendon elongation | 2 months
  The difference (mm) between the calculated length changes of the muscle-tendon unit and the muscle-length changes recorded by the ultrasound.
Achilles tendon stiffness | 2 months
  The achilles tendon stiffness (N/m) was calculated through linear regression of the absolute tendon force and related changes in tendon length.
Achilles tendon strain | 2 months
  The achilles tendon strain (%) was calculated as the tendon elongation divided by the initial tendon length
Achilles tendon stress | 2 months
  The achilles tendon stress was calculated as the tendon elongation divided by the initial tendon length and expressed in (N/mm2).
Young's modulus | 2 months
  Young's modulus (N/mm2) was calculated as the ratio of achilles tendon tensile stress to tensile strain

CONTACTS AND LOCATIONS:
Overall Officials: Ragab K Elnaggar, PhD, Principal Investigator — Prince Sattam Bin Abdulaziz University
Locations (1):
- Ragab K. Elnaggar, Al Kharj, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No